CLINICAL TRIAL: NCT02719184
Title: Observational Study in Healthy Subjects and Patients With COPD to Assess the Relationship Between Clinical, Imaging and Biomarker Measurements, and Progression of Emphysema Over Three Years [FOOTPRINTS®].
Brief Title: Longitudinal Follow up to Assess Biomarkers Predictive of Emphysema Progression in Patients With COPD (Chronic Obstructive Pulmonary Disease)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 352.2069
Record Dates: First submitted 2016-03-18; First posted 2016-03-25 (Estimated); Results first posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Pulmonary Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Soluble and imaging biomarkers

GROUPS / COHORTS (5):
- Healthy subjects: All eligible healthy subjects were included in this group. The observational period is 156 weeks.
- COPD GOLD I: All eligible patients with Chronic Obstructive Pulmonary Disease (COPD) grade 1 according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) were included in this group. The observational period is 156 weeks.
- COPD GOLD II: All eligible patients with Chronic Obstructive Pulmonary Disease (COPD) grade 2 according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) were included in this group. The observational period is 156 weeks.
- COPD GOLD III: All eligible patients with Chronic Obstructive Pulmonary Disease (COPD) grade 3 according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) were included in this group. The observational period is 156 weeks.
- COPD and A1AT Deficiency: All eligible patients with Chronic Obstructive Pulmonary Disease (COPD) and Alpha one anti-trypsin (A1AT) deficiency were included in this group. The observational period is 156 weeks.

SUMMARY:
The study will include 60 healthy subjects (ex-smoker without any airflow limitation), 125 COPD GOLD (global initiative for chronic obstructive lung disease) I , 125 COPD GOLD II, 125 COPD GOLD III and up to 20 patients with COPD and A1AT (Alpha1-Antitrypsin) deficiency (ZZ genotype). Soluble and imaging biomarkers will be investigated addressing different aspects of disease pathways postulated to be relevant for COPD progression.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

* Male or female healthy subjects or COPD (GOLD I to III) outpatients with or without A1AT deficiency
* Ex-smokers for at least 9 months with a smoking history of >=20 pack years
* Signed informed consent consistent with ICH-GCP (International Conference on Harmonisation - Good Clinical Practice) guidelines prior to participation in the study, which includes the application of study restrictions
* Age >= 40 and <=70 years
* Body mass index (BMI) of >= 18 and <= 35 kg/m2 (<= 30 kg/m2 in the MRI subset)
* Ability to perform all study related procedures including technically acceptable pulmonary function tests, body plethysmography, DLCO ( Diffusing Capacity of the lungs for Carbon Monoxide) , sputum induction (if applicable), chest CT (Computed Tomography) and MRI (if applicable)

Inclusion Criteria Specific for Patients with COPD - Patients must have a current diagnosis of COPD made by a physician prior to or during Visit 1 and a mMRC (Modified Medical Research Council Dyspnea Scale) score of 1 or more. The diagnosis of COPD must be in accordance with GOLD Guidelines and must be documented by the following criteria: Known relatively stable airway obstruction with a post-bronchodilator FEV1 (Forced Expiratory Volume in first second)/FVC (Forced Vital Capacity) < 70 %

* The current COPD must be mild, moderate or severe based on lung functions and symptoms and the clinical situation must have stabilized for at least 4 weeks prior to Visit 1. The following definitions adapted from the GOLD Guidelines apply:

  1. mild: post-broncho-dilator FEV1 >=80% of predicted normal (GLI 2012 and JRS 2014) at Visit 1
  2. moderate: 50%<= post-broncho-dilator FEV1 < 80% of predicted normal (GLI 2012 and JRS 2014) without chronic respiratory failure at Visit 1
  3. severe: 30%<= post-bronchodilator FEV1 <50% of predicted normal (GLI 2012 and JRS 2014) without chronic respiratory failure at Visit 1
* Patients must be on stable therapy (not limited to respiratory medication) for the last 4 weeks prior to Visit 1

Inclusion Criteria Specific Patients with COPD and A1AT Deficiency

- Documented A1AT deficiency of ZZ genotype

Inclusion Criteria Specific Healthy Subjects

* Normal lung function values at Visit 1 with a documented post-bronchodilator FEV1 >=80% of predicted normal (GLI 2012 and JRS 2014) and a post-bronchodilator FEV1/FVC >= lower limit of normal
* Mean post DLCO over all acceptable measurements at Visit 1 of >= 70% of predicted normal
* Further inclusion criteria apply

Exclusion Criteria:

General Exclusion Criteria

* Previous participation in this study or participation in another trial with an investigational drug within 6 weeks prior to Visit 1 or during the study
* Significant pulmonary disease or other significant medical conditions* (as determined by medical history, examination and clinical investigations at screening) that may in the opinion of the investigator result in any of the following:

  1. Put the subject at risk because of participation in the study
  2. Cause concern regarding the subject's ability to participate in this study *e.g. rheumatoid arthritis, inflammatory bowel disease, severe liver disease, psoriasis, hematological, infectious and psychiatric diseases
* Documented history of asthma. For allergic rhinitis or atopy, source documentation to verify that the subject does not have asthma
* Planned surgery during the study expected to interfere with study procedures and outcome
* Blood withdrawal of more than 100 mL within the past 6 weeks prior to Visit 1 and between Visit 1 and 2
* Significant alcohol or drug abuse within past 2 years prior to Visit 1
* Women who are pregnant, nursing or plan to become pregnant while in the study
* Place of permanent residence of less than 3 months prior to Visit 1
* For the MRI subset: subject who do not meet the following criteria for the MRI assessment at Visit 2: systolic blood pressure between 90 and 180 mmHg (SBP), diastolic blood pressure between 50 and 110 mmHg (DBP), pulse rate between 40 and 110 bpm, ear temperature between 35 - 37.5 C, and a glomerular filtration rate (GFR) >= 30 mL/min (GFR must not be older than 14 days from the MRI assessment)

Exclusion Criteria Specific for Patients with COPD

- Respiratory tract infection or COPD exacerbation in the 4 weeks prior to Visit 1 or during the screening period prior to Visit 2, if rescheduling rules cannot be met

Exclusion Criteria Specific Patients with COPD and A1AT Deficiency

* Newly added anti-inflammatory treatment within 4 weeks prior to Visit 1
* Patients on treatment with PDE (Phosphodiesterase)-5 inhibitors (e.g. Roflumilast) and maintenance treatment Methylxanthines (e.g. Theophylline)
* Hospitalisation for respiratory failure during the year prior to Visit 1
* A history of cystic fibrosis
* Clinical diagnosis of bronchiectasis requiring specific treatment
* Clinically relevant abnormal baseline hematology and blood chemistry
* Known active tuberculosis
* Patients with change in any therapy within 4 weeks prior to Visit 1
* Current and planned A1AT augmentation therapy
* A malignancy for which the patient has undergone resection, radiation or chemotherapy within past 5 years. Patients with treated basal cell carcinoma or fully cured squamous cell carcinoma are allowed
* Inability to comply with restrictions regarding diet, life style and medication
* Further exclusion criteria apply

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers and COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (51):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Diego, San Diego, California
  - The Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - National Jewish Health, Denver, Colorado
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
- Belgium (2):
  - Brussels - UNIV St-Pierre, Brussels
  - UZ Leuven, Leuven
- Canada (6):
  - University of Alberta Hospital (University of Alberta), Edmonton, Alberta
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
  - IUCPQ (Laval University), Québec
- Denmark (3):
  - Aarhus University Hospital, Aarhus N
  - Gentofte Hospital, Hellerup
  - Hvidovre Hospital, Hvidovre
- Finland (2):
  - HYKS Keuhkosairauksien tutkimusyksikkö, Helsinki
  - TYKS, Turku
- Germany (4):
  - IKF Pneumologie GmbH & Co. KG, Frankfurt
  - Pneumologisches Forschungsinstitut an der LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Fraunhofer ITEM, Hanover
  - KLB Gesundheitsforschung Lübeck GmbH, Lübeck
- Japan (5):
  - Kagoshima University Hospital, Kagoshima, Kagoshima
  - Showa University Fujigaoka Hospital, Kanagawa, Yokohama
  - Kishiwada City Hospital, Osaka, Kishiwada
  - Osaka City University Hospital, Osaka, Osaka
  - Showa University Hospital, Tokyo, Shinagawa-ku
- Poland (3):
  - Respiratory Medicine Centre, private prac., Bialystok, Bialystok
  - University Clinical Center, Gdansk, Gdansk
  - Institute of Tuberculosis & Lung Disease, Warsaw, Warsaw
- South Korea (4):
  - Konkuk University Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
- Spain (6):
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Quirónsalud Madrid, Pozuelo de Alarcón
- Skånes universitetssjukhus, Lund, Lund, Sweden
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - Glenfield Hospital, Leicester
  - Royal Free Hospital, London
  - Medicines Evaluation Unit, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Crapo JD, Gupta A, Lynch DA, Turner AM, Mroz RM, Janssens W, Ludwig-Sengpiel A, Koegler H, Eleftheraki A, Risse F, Diefenbach C. Baseline characteristics from a 3-year longitudinal study to phenotype subjects with COPD: the FOOTPRINTS study. Respir Res. 2023 Nov 17;24(1):290. doi: 10.1186/s12931-023-02584-2. PMID 37978492
- [Derived] Crapo J, Gupta A, Lynch DA, Vogel-Claussen J, Watz H, Turner AM, Mroz RM, Janssens W, Ludwig-Sengpiel A, Beck M, Langellier B, Ittrich C, Risse F, Diefenbach C. FOOTPRINTS study protocol: rationale and methodology of a 3-year longitudinal observational study to phenotype patients with COPD. BMJ Open. 2021 Mar 22;11(3):e042526. doi: 10.1136/bmjopen-2020-042526. PMID 33753437
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The overall objective of this study is to explore, if any of the biomarkers (soluble, functional imaging and physiological) assessed within healthy subjects, patients with Chronic Obstructive Pulmonary Disease (COPD) and patients with COPD and Alpha-1 Antitrypsin (A1AT) deficiency are correlated to COPD disease progression, particularly emphysema progression over 156 weeks.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
Period: Overall Study
Arm/Group | Healthy Subjects | COPD GOLD I | COPD GOLD II | COPD GOLD III | COPD and A1AT Deficiency
Started ("Started" = Observed subjects set) | 62 | 123 | 130 | 129 | 19
Per-Protocol Set (Biomarker Subjects) | 61 | 122 | 127 | 127 | 19
Completed | 56 | 101 | 110 | 93 | 10
Not Completed | 6 | 22 | 20 | 36 | 9
Not completed — Other than listed | 1 | 12 | 13 | 22 | 9
Not completed — Withdrawal by Subject | 5 | 3 | 6 | 6 | 0
Not completed — Lost to Follow-up | 0 | 4 | 1 | 3 | 0
Not completed — Protocol Violation | 0 | 3 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Observed subjects set (OBS): All subjects, from the Screened subjects set (SCR), who are eligible to enter the observation period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Subjects | COPD GOLD I | COPD GOLD II | COPD GOLD III | COPD and A1AT Deficiency | Total
Number analyzed (Participants) | 62 | 123 | 130 | 129 | 19 | 463
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.0 (6.8) | 61.9 (6.2) | 61.8 (5.3) | 62.9 (5.6) | 52.8 (9.0) | 60.7 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 37 | 52 | 49 | 3 | 164
  Male | 39 | 86 | 78 | 80 | 16 | 299
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 3 | 1 | 7
  Not Hispanic or Latino | 61 | 121 | 127 | 124 | 18 | 451
  Unknown or Not Reported | 1 | 0 | 2 | 2 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 0 | 2
  Asian | 8 | 16 | 7 | 6 | 0 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 4 | 3 | 0 | 10
  White | 52 | 106 | 117 | 119 | 19 | 413
  More than one race | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 00 | 0 | 0
Adjusted lung density (ALD) [Mean (Standard Deviation); unit: gram/Liter] — The ALD was calculated as: Percentile Density at 15% (PD15) [gram/Liter (L)] * (Inspiratory volume [L]/predicted total lung volume [L]). Population: Per-Protocol Set (Biomarker Subjects): All subjects, from the Observed subjects set, who have no Important Protocol Deviations (IPDs) affecting the clinical or biomarker assessments.
  gram/Liter
    number analyzed (Participants) | 55 | 100 | 89 | 89 | 13 | 346
    (all) | 88.50 (13.90) | 86.20 (21.38) | 72.42 (21.69) | 54.81 (23.08) | 50.86 (18.15) | 73.62 (24.92)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline at Week 156 in Adjusted Lung Density (ALD) Based on Percentile Density at 15% (PD15) Adjusted for Lung Volume
Description: The absolute change from baseline at Week 156 in adjusted lung density (ALD) based on Percentile Density at 15% (PD15) adjusted for lung volume was reported. The ALD was calculated as: Percentile Density at 15% (PD15) [gram/Liter (L)] * (Inspiratory volume [L]/predicted total lung volume [L]). The absolute change from baseline in ALD gram/Liter (g/L) was analyzed by Mixed Model for Repeated Measures (MMRM).
Time Frame: Up to Week 156. Change from baseline value at Week 156 was reported.
Population: Per-Protocol Set (Biomarker Subjects): All subjects, from the Observed subjects set, who have no Important Protocol Deviations (IPDs) affecting the clinical or biomarker assessments. Only participants with non-missing results were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: gram/Liter (g/L)
Arm/Group | Healthy Subjects | COPD GOLD I | COPD GOLD II | COPD GOLD III | COPD and A1AT Deficiency
Number analyzed (Participants) | 41 | 64 | 51 | 37 | 5
gram/Liter (g/L) | -0.27 (1.00) | -3.15 (0.79) | -5.04 (0.84) | -4.74 (1.04) | -6.13 (2.51)
Statistical Analysis 1: Comparison: Healthy Subjects vs COPD GOLD I; Test type: Other — The analysis was based on a Mixed Model for Repeated Measures (MMRM) approach with diagnosis group-by-visit and baseline ALD value-by-visit terms, and unstructured covariance matrix structure for repeated measurements within subject; p = 0.0202, Mixed Model for Repeated Measures (MMRM); Adjusted mean difference = -2.89, 95% CI 2-sided [-5.32 to -0.45], Standard Error of Mean 1.23 — The mean difference was calculated as value from COPD GOLD I group - value from Healthy subjects group
Statistical Analysis 2: Comparison: Healthy Subjects vs COPD GOLD II; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0003, Mixed Model for Repeated Measures (MMRM); Adjusted mean difference = -4.78, 95% CI 2-sided [-7.36 to -2.19], Standard Error of Mean 1.31 — The mean difference was calculated as value from COPD GOLD II group - value from Healthy subjects group
Statistical Analysis 3: Comparison: Healthy Subjects vs COPD GOLD III; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0033, Mixed Model for Repeated Measures (MMRM); Adjusted mean difference = -4.47, 95% CI 2-sided [-7.44 to -1.50], Standard Error of Mean 1.51 — The mean difference was calculated as value from COPD GOLD III group - value from Healthy subjects group
Statistical Analysis 4: Comparison: Healthy Subjects vs COPD and A1AT Deficiency; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0334, Mixed Model for Repeated Measures (MMRM); Adjusted mean difference = -5.86, 95% CI 2-sided [-11.26 to -0.47], Standard Error of Mean 2.74 — The mean difference was calculated as value from COPD and A1AT group - value from Healthy subjects group

2. Primary Outcome: Annual Rate of Lung Function Decline Based on Forced Expiratory Volume in 1 Second (FEV1)
Description: The annual rate of lung function decline based on Forced Expiratory Volume in 1 second (FEV1) was reported. The annual rate was estimated from a random slope and intercept model with fixed categorical effects of diagnosis group, fixed continuous effects of time [Year], and including diagnosis group-by-time interaction. Random effect was included for subject specific intercept and time. Within-subject errors are modelled by an unstructured variance-covariance matrix.
Time Frame: Up to Week 156
Population: as for outcome 1
Measure: Mean (Standard Error); unit: milliliter / year [mL/year]
Arm/Group | Healthy Subjects | COPD GOLD I | COPD GOLD II | COPD GOLD III | COPD and A1AT Deficiency
Number analyzed (Participants) | 55 | 106 | 101 | 90 | 14
milliliter / year [mL/year] | -25.7 (11.4) | -24.4 (8.9) | -44.9 (9.6) | -59.3 (11.4) | -87.5 (28.0)
Statistical Analysis 1: Comparison: Healthy Subjects vs COPD GOLD I; Test type: Other — A random slope and intercept model with fixed categorical effects of diagnosis group, fixed continuous effects of time, and including diagnosis group-by-time interaction was applied. Random effect was included for subject specific intercept and time. Within-subject errors are modelled by an unstructured variance-covariance matrix; p = 0.9306, Random slope and intercept model; Unadjusted mean difference = 1.3, 95% CI 2-sided [-27.2 to 29.7], Standard Error of Mean 14.4 — The mean difference was calculated as value from COPD GOLD I group - value from Healthy subjects group
Statistical Analysis 2: Comparison: Healthy Subjects vs COPD GOLD II; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.1983, Random slope and intercept model; The mean difference was calculated as value from COPD GOLD II group - value from Healthy subjects group; Unadjusted mean difference = -19.2, 95% CI 2-sided [-48.5 to 10.1], Standard Error of Mean 14.9
Statistical Analysis 3: Comparison: Healthy Subjects vs COPD GOLD III; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0381, Random slope and intercept model; Unadjusted mean difference = -33.6, 95% CI 2-sided [-65.4 to -1.9], Standard Error of Mean 16.1 — The mean difference was calculated as value from COPD GOLD III group - value from Healthy subjects group
Statistical Analysis 4: Comparison: Healthy Subjects vs COPD and A1AT Deficiency; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0419, Random slope and intercept model; Unadjusted mean difference = -61.8, 95% CI 2-sided [-121.3 to -2.3], Standard Error of Mean 30.3 — The mean difference was calculated as value from COPD and A1AT group - value from Healthy subjects group

3. Primary Outcome: Number of Participants by the Category of Number of Exacerbations During Study
Description: Number of participants by the category of number of exacerbations (no exacerbation, 1 exacerbation, or >= 2 exacerbations) during study was reported.
Time Frame: Up to Week 156
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Subjects | COPD GOLD I | COPD GOLD II | COPD GOLD III | COPD and A1AT Deficiency
Number analyzed (Participants) | 61 | 122 | 127 | 127 | 19
Participants
  0 | 59 | 89 | 66 | 41 | 2
  1 | 1 | 23 | 24 | 30 | 4
  >= 2 | 1 | 10 | 37 | 56 | 13

4. Primary Outcome: Duration of Exacerbations During Study (Per Year)
Description: The duration of exacerbations for each subject was calculated as: sum of duration of episodes during study (days)*(365.25/ number of days in study).
Time Frame: Up to 156 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days/year
Arm/Group | Healthy Subjects | COPD GOLD I | COPD GOLD II | COPD GOLD III | COPD and A1AT Deficiency
Number analyzed (Participants) | 2 | 33 | 61 | 86 | 17
days/year | 13.1 (5.2) | 9.7 (13.0) | 18.0 (19.4) | 19.7 (24.2) | 17.8 (16.7)

5. Primary Outcome: Number of Participants With at Least Moderate Exacerbation During Study by the Category of Number of Moderate Exacerbations
Description: Number of participants with at least moderate exacerbation during study by the category of number of moderate exacerbation (no moderate exacerbation, 1 moderate exacerbation, or >= 2 moderate exacerbations) was reported.
Time Frame: Up to 156 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Subjects | COPD GOLD I | COPD GOLD II | COPD GOLD III | COPD and A1AT Deficiency
Number analyzed (Participants) | 61 | 122 | 127 | 127 | 19
Participants
  0 | 60 | 93 | 73 | 48 | 4
  1 | 1 | 20 | 22 | 29 | 8
  >= 2 | 0 | 9 | 32 | 50 | 7

6. Primary Outcome: Number of Participants With Severe Exacerbations During Study by the Category of Number of Severe Exacerbations
Description: Number of participants with severe exacerbations during study by the category of number of severe exacerbations (no severe exacerbation, 1 severe exacerbation, or >= 2 severe exacerbations) was reported.
Time Frame: Up to 156 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Subjects | COPD GOLD I | COPD GOLD II | COPD GOLD III | COPD and A1AT Deficiency
Number analyzed (Participants) | 61 | 122 | 127 | 127 | 19
Participants
  0 | 61 | 120 | 118 | 103 | 16
  1 | 0 | 1 | 9 | 19 | 1
  >= 2 | 0 | 1 | 0 | 5 | 2

ADVERSE EVENTS:
Time Frame: From Day 1 of the study until end of observational period, up to 156 weeks.
Description: Observed subjects set (OBS): All subjects, from the Screened subjects set (SCR), who are eligible to enter the observation period. Only procedure related adverse events were collected and reported for this study.
Arm/Group | Healthy Subjects | COPD GOLD I | COPD GOLD II | COPD GOLD III | COPD and A1AT Deficiency
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/123 | 0/130 | 0/129 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/123 | 0/130 | 0/129 | 0/19
Other Adverse Events (participants affected / at risk) | 0/62 | 0/123 | 0/130 | 0/129 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT02719184/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT02719184/SAP_001.pdf